CLINICAL TRIAL: NCT02055651
Title: Descriptive Observational Study of Cardiovascular Health Risk Factors in Workers of Bayer S.A. Company in São Paulo
Brief Title: Cardiovascular Disease Risk Factors Prevalence Among Bayer's Employees in São Paulo, Brazil
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17312; NN1325BR (Other: Company internal)
Record Dates: First submitted 2014-01-24; First posted 2014-02-05 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Occupational Health
Keywords: Worksite; Cardiovascular; Epidemiology; Risk factors
MeSH Terms: interventions — Restraint, Physical; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bayer Sao Paulo employees: Workers from Bayer in site Socorro who participate in the trial
  Interventions: Behavioral: Examination and survey

INTERVENTIONS:
Behavioral: Examination and survey — Routine medical examination as required by law and follow-up for lifestyle change program

SUMMARY:
Introduction: As employees spent most part of their time at the worksite, it provides a venue to address multiple individual risk factors and promote health. The America Heart Association (AHA) defined cardiovascular health using as metrics smoking status, body mass index, physical activity, diet, total cholesterol, blood pressure and fasting blood glucose.

Objective: Evaluate Bayer employees' cardiovascular health according to the AHA definition and the acceptance to engage in lifestyle change programs.

Methods: By the time of the annual occupational safety periodic medical examination, employees will receive an email with information about the cardiovascular health screening, exams requisition (fasting blood glucose and total cholesterol) and a copy of the written informed consent. If the employee accepts to participate, after providing a written informed consent, he will be evaluated according to the AHA cardiovascular health metrics. Data will be collected at the occupational safety electronic health record. After medical evaluation, employees will receive a printed feedback with their cardiovascular health score and will be referred to indicated lifestyle change programs (healthy weight, smoking cessation, diabetes control, high blood pressure control, dyslipidemia control).

After 12 months we will evaluate the percentage of employees who accept to participate; prevalence of the cardiovascular risk factors and distribution according to the AHA classification in ideal, intermediate and poor; adherence to lifestyle change programs.

ELIGIBILITY:
Inclusion Criteria:

* Employees with 20 years of age or more that daily work at Bayer's site in São Paulo
* Provide written informed consent

Exclusion Criteria:

* Employees that will no longer work for Bayer in 30 days
* Employees that are retired from work during the study period

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bayer's employees (São Paulo, Brazil)
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Cardiovascular health metrics on a three-point scale (poor, intermediate, ideal) | 1 day
  Metrics are defined by the American Heart Association (AHA) [Lloyd-Jones and cols, 2010]

SECONDARY OUTCOMES:
Number of participants who are suggested to participate in a lifestyle change program and show up for at least one session | Up to 4 weeks after cardiovascular examination

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- São Paulo, Brazil